CLINICAL TRIAL: NCT03251105
Title: Comparison of the Supreme™ And Proseal™ Laryngeal Mask Airways in Infants: A Prospective Randomised Clinical Study
Brief Title: Supreme Versus Proseal Laryngeal Mask Airways in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Canan Tulay ISIL, Specialist, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEEAH/26.04.2016/659
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Surgery; Infant Conditions; Anesthesia

STUDY DESIGN:
Intervention Model Description: Infants, who were scheduled to undergo lower abdominal surgery and to receive anaesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProSeal group (Active Comparator): This group received the ProSeal LMA for supraglottic airway intubation and ventilation during anaesthesia.
  Interventions: Device: supraglottic airway intubation
- Supreme group (Active Comparator): This group received the Supreme LMA for supraglottic airway intubation and ventilation during anaesthesia.
  Interventions: Device: supraglottic airway intubation

INTERVENTIONS:
Device: supraglottic airway intubation

SUMMARY:
In this study, the Supreme and ProSeal LMAs in infants were compared by measuring their performance characteristics, including insertion features, ventilation parameters, induced changes in hemodynamics and rates of postoperative complications.

DETAILED DESCRIPTION:
Both the Supreme™ and ProSeal™ laryngeal mask airways (LMAs) are widely used for paediatric anaesthesia; however, LMA use in infants is limited, as many anaesthesiologists prefer to use tracheal intubation in infants.

In this study, the Supreme and ProSeal LMAs in infants were compared by measuring their performance characteristics, including insertion features, ventilation parameters, induced changes in hemodynamics and rates of postoperative complications.

Infants of ASA physical status I who were scheduled for elective, minor, lower abdominal surgery were divided into two groups: the Supreme LMA group and the ProSeal LMA group. Heart rate (HR), oxygen saturation and end tidal carbon dioxide values were recorded both before and after LMA insertion, as well as both before and after extubation. After extubation, complications and adverse effects were noted.

Demographics and surgical data were similar between the two groups. LMA insertion times for the ProSeal group were shorter, the leakage pressure for the ProSeal group was statistically higher. The ProSeal LMA is superior to the Supreme LMA for use in infants, due to its ease of insertion, high oropharyngeal leakage pressure and fewer induced changes in hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective, minor (<1 hour duration), lower abdominal surgery, including unilateral herniorrhaphy and unilateral orchidopexy

Exclusion Criteria:

* premature birth, potentially difficult airway, clinically significant upper respiratory tract infection and risk of aspiration, such as gastro-oesophageal reflux disease

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
performance characteristics | operation duration
  insertion time in minutes

SECONDARY OUTCOMES:
haemodynamics | operation duration
  end tidal CO2 (EtCO2) in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Oba, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
We can only share data as Exel or SSPS, but not with patient names.

REFERENCES:
- [Background] Luce V, Harkouk H, Brasher C, Michelet D, Hilly J, Maesani M, Diallo T, Mangalsuren N, Nivoche Y, Dahmani S. Supraglottic airway devices vs tracheal intubation in children: a quantitative meta-analysis of respiratory complications. Paediatr Anaesth. 2014 Oct;24(10):1088-98. doi: 10.1111/pan.12495. Epub 2014 Jul 30. PMID 25074619
- [Derived] Oba S, Turk HS, Isil CT, Erdogan H, Sayin P, Dokucu AI. Comparison of the Supreme and ProSeal laryngeal mask airways in infants: a prospective randomised clinical study. BMC Anesthesiol. 2017 Sep 5;17(1):125. doi: 10.1186/s12871-017-0418-z. PMID 28870163